CLINICAL TRIAL: NCT01788124
Title: A Randomized Prospective Trial Comparing Metal to Plastic Speculums for Patient Comfort
Brief Title: A Prospective Trial Comparing Metal to Plastic Speculums for Patient Comfort
Acronym: GYN
Status: Completed | Type: Observational
Sponsor: St. John Health System, Michigan (Other)
Responsible Party: Principal Investigator, Michael Shaw PhD, Research Coordinator, St. John Health System, Michigan
Other Study IDs: macomb0001
Record Dates: First submitted 2013-02-04; First posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Patient Comfort
Keywords: Speculum; Metal; Plastic; Visual Analoge Scale; Discomfort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Metal Speculum: exam with metal speculum
- Plastic Speculum: exam with plastic speculum

SUMMARY:
The purpose of this study is to evaluate the comfort of two type of speculums used during routine gynecologic exam. Your treatment and medical care will not change because you are participating in this study. Your doctor will continue to make all decisions regarding your proper treatment and care.

DETAILED DESCRIPTION:
Speculum examination is a common procedure in the gynecology clinic used for evaluation of numerous conditions such as vaginitis, and during cervical cytology screening (PAP smears). The speculum is inserted into the woman's vagina and used to keep the vaginal walls apart during exam and procedures. Each step of the examination with a speculum including insertion, manipulation during examination, and removal can cause discomfort for the patient. Fear of examination pain is considered one barrier to examination compliance. Any method to decrease discomfort during the exam would be considered beneficial to patient screening.

Typically two types of speculums are used in clinical practice, metal and plastic. There are advantages to both, and usage is usually predicated by physician preference. Previous studies have demonstrated a clear difference in patient comfort between metal speculums and newer dilating speculums such as the Vera scope (1). Clinical trials have also shown the benefit of using lubrication on metal speculums during routine exams (2). To date there are no clinical trails to examine the difference in patient comfort between metal and plastic bi-valve speculums.

ELIGIBILITY:
Inclusion Criteria:

* Any woman presenting to Great Lakes Obstetrics and Gynecology or Macomb Academic OB/GYN Clinic for a routine gynecological exam
* Women ≥ 18 years of age
* Women willing and able to give informed consent according to the guidelines established by the St John IRB

Exclusion Criteria:

* Patients that can not or will not sign the informed consent document
* Women whose English language skills are insufficient to understand the written informed consent or the post examination questionnaire.
* Any woman for who use of a speculum is contraindicated.
* Any woman with a condition that might alter pain perception
* Current pain medication use
* History of drug abuse
* History of painful speculum examination
* Menopausal women
* Women who are pregnant or within 6 weeks of delivery
* Women presenting with dyspareunia, vaginitis, vulvar pain or vulvar lesions
* Women presenting for a vulvar, vaginal or uterine procedure.
* Women who have had a previous abnormal PAP smear (Cervical Intraepithelial Neoplasia >1)
* Women ≤ 18 years of age.
* Women who have never had vaginal intercourse.
* Women who have never had a speculum examination in the past

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women greater than 18 years of age presenting for routine speculum exam
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Patient Discomfort VAS | up to one day post exam
  . Patients presenting for routine gynecological examination will be randomized to either plastic or metal speculum arm. Patient discomfort will be assessed using a self administered visual analogue scale (VAS). Patient comfort between groups will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- St John Macomb Oakland Hospital, Warren, Michigan, United States